CLINICAL TRIAL: NCT05509335
Title: Ultrasound Assessment On Real Time Effectiveness Of Cricoid Pressure In Paediatric Population Under General Anaesthesia
Brief Title: Ultrasound Assessment On Effectiveness of Cricoid Pressure In Paediatric Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr. Cheong Chao Chia, Clinical Anaesthesiologist, Lecturer, University of Malaya
Other Study IDs: 2021329-9999
Record Dates: First submitted 2022-08-14; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Aspiration of Food; Pediatric ALL
Keywords: cricoid pressure; oesophagus position; pediatric
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cricoid pressure (CP) confers Grade IIA evidence in preventing gastric insufflation during general anaesthesia. However, a retrospective review of computed tomography scans by Dotson et al. shows that 45% oesophagus is eccentric in the paediatric population aged 1 to 8 years old. In adults, the eccentric oesophagus is associated with reduced CP efficacy in occluding oesophagus. To date, no dynamic real-time study has been done to assess the incidence of the eccentric oesophagus in the paediatric population, the efficacy of CP in occluding eccentric oesophagus, and the effect of anaesthesia on oesophageal position.

Any patients aged 1 to 8 years old are eligible to participate This study will be conducted in the operation theatre of UMMC. The investigators plan to perform an ultrasound of the neck throughout the phases of anaesthetic induction and determine the oesophagus position and its compressibility with CP application.

DETAILED DESCRIPTION:
In a survey presented by Society for Paediatric Anaesthesia in 2004, 68% of paediatric anaesthesiologists apply CP to prevent passive regurgitation of food into the pharynx. 33% of respondents use CP to prevent gastric insufflation during mask ventilation. Among the respondent, only 24% responded CP reliably occludes the oesophageal lumen.

The anatomically central oesophagus lies behind cricoid cartilage, by applying CP oesophageal lumen will be occluded. However, it remains debatable if eccentric oesophageal is compressible. Studies were conducted on the adult population. Efficacy of CP has been studied in adult patients by means of magnetic resonance imaging. It was shown that CP was ineffective in occluding the oesophageal lumen in adult patients with an eccentric oesophagus. In addition, the study raised the concern of CP application in itself might result in lateral displacement of the oesophagus. This is further supported by Lim et al.'s study which shows the ineffectiveness of CP in occluding eccentric oesophagus in adult patients.

Contrary to the aforementioned studies, Rice et al's demonstrated oesophagus was occludable regardless of the position. The author hypothesized that the hypopharynx and cricoid move as one anatomical unit and the oesophagus would be compressed following the application of CP.

Although the effectiveness of CP was extensively studied in the adult population, studies on the paediatric population remained scarce. A retrospective review of computed tomography scans by Dotson et al. shows that 45% oesophagus is eccentric in the paediatric population aged 1 to 8 years old. In our pilot study, the investigators found out that 90 per cent of the oesophagus in the paediatric population was successfully occluded following the application of CP regardless of its position.

Cricoid pressure is not without risk. CP was associated with oesophageal rupture. It has been known to disrupt the laryngoscopic view of the glottis and cause difficult intubation. Hence, it would be imperative to investigate whether CP is truly effective in occluding the oesophagus and preventing gastric aspiration in the paediatric population.

This would be a prospective observational study to study the real-time dynamic effect of oesophageal position and the effect of anaesthesia on oesophageal position. Most importantly, the investigators are hoping to investigate the effectiveness of CP in occluding oesophagus in the paediatric population.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1, 2
* Age 1-8 years old
* Scheduled for surgery under general anaesthesia requiring tracheal intubation

Exclusion Criteria:

* Presence of neck mass/ cervical spine pathology, prior neck surgery
* Pathology of the upper respiratory tract
* Anticipated difficult intubation / difficult mask ventilation
* Risk of pulmonary aspiration of gastric contents (eg. Gastroesophageal reflux disease, hiatus hernia, intestinal obstruction)
* Morbid obesity BMI ≥ 35 kg/m2 (above 85th centile) - overweight patients
* Inadequate fasting ( 6 hours solid food/ formula milk, 4 hours breast milk and 2 hours clear fluid) - definite indication for rapid sequence induction
* Uncontrolled cardiopulmonary disease
* Oesophageal conditions: achalasia, Zenker's diverticulum

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: ASA 1 and 2 children aged 1 to 8 years old undergoing general anaesthesia for elective surgery requires muscle paralysis and tracheal intubation. We rule out cases which need rapid sequence induction, high risk of aspiration and difficult airway.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-08-19 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of oesophagus compressible following application of CP in paediatric population | Through study completion, average 1 year
  A published study quoted 45% lateral displacement of the oesophagus in younger children, the incidence was derived from a retrospective review of CT neck in children. Eccentric oesophagus has been associated with ineffective CP in adults. The investigators use ultrasound to determine the location of the oesophagus relative to the trachea. If the oesophagus is central, we assume CP is effective. On the other hand, if the oesophagus is eccentric, ultrasound would be used to assess the compressibility of the oesophagus following CP.

SECONDARY OUTCOMES:
Determine incidence of eccentric oesophagus in paediatric population under effect of general anaesthesia | Through study completion, average 1 year
  A published study was conducted from a retrospective review of CT cervical spine of children which found 45% eccentric oesophagus in younger children. However, the position was determined in awake patients with no effect of the anaesthetic drug. We like to investigate the effect of general anaesthetic agents (in particular muscle relaxant) on oesophagus position.
Determine incidence of lateral displacement of oesophagus during CP | Through study completion, average 1 year
  From our pilot study on 10 children aged < 8 years old, we observed centrally located oesophagus was displaced following the application of CP. We would like to investigate the incidence of this phenomenon and if there is a shift of oesophageal position, would the application of CP be effective in occluding the oesophagus.

CONTACTS AND LOCATIONS:
Overall Officials: Chew Yin Wang, FRCA, Study Chair — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
result and data

REFERENCES:
- [Background] Dotson K, Kiger J, Carpenter C, Lewis M, Hill J, Raney L, Losek JD. Alignment of cricoid cartilage and esophagus and its potential influence on the effectiveness of Sellick maneuver in children. Pediatr Emerg Care. 2010 Oct;26(10):722-5. doi: 10.1097/PEC.0b013e3181f39b74. PMID 20881908
- [Background] Andruszkiewicz P, Wojtczak J, Wroblewski L, Kaczor M, Sobczyk D, Kowalik I. Ultrasound evaluation of the impact of cricoid pressure versus novel 'paralaryngeal pressure' on anteroposterior oesophageal diameter. Anaesthesia. 2016 Sep;71(9):1024-9. doi: 10.1111/anae.13518. PMID 27523050
- [Background] Birenbaum A, Hajage D, Roche S, Ntouba A, Eurin M, Cuvillon P, Rohn A, Compere V, Benhamou D, Biais M, Menut R, Benachi S, Lenfant F, Riou B; IRIS Investigators Group. Effect of Cricoid Pressure Compared With a Sham Procedure in the Rapid Sequence Induction of Anesthesia: The IRIS Randomized Clinical Trial. JAMA Surg. 2019 Jan 1;154(1):9-17. doi: 10.1001/jamasurg.2018.3577. PMID 30347104
- [Background] Boet S, Duttchen K, Chan J, Chan AW, Morrish W, Ferland A, Hare GM, Hong AP. Cricoid pressure provides incomplete esophageal occlusion associated with lateral deviation: a magnetic resonance imaging study. J Emerg Med. 2012 May;42(5):606-11. doi: 10.1016/j.jemermed.2011.05.014. Epub 2011 Jun 12. PMID 21669510